CLINICAL TRIAL: NCT06044389
Title: Anwendungsbeobachtung Zur Sicherheit Und Wirkung Des Medizinproduktes Fructosin®
Brief Title: Observational Study on the Safety and Efficacy of the Medical Product Fructosin.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sciotec Diagnostic Technologies GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: BTS1295/18
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Fructose Intolerance
MeSH Terms: conditions — Fructose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People suffering from fructose intolerance
  Interventions: Device: Fructosin

INTERVENTIONS:
Device: Fructosin — Fructosin® is a CE marked medical device. The capsules with 30.23 mg xylose isomerase are taken as recommended. This means that, depending on the total intake, 1-2 capsules are to be taken with water 15 minutes before meals containing fructose, a maximum of 3 times a day.
  Use as needed during the 4-week intake phase.
  Other Names: Fructease

SUMMARY:
Fructosin® is a medical device for use in fructose intolerance. In this uncontrolled posdt market clinical follow up (PMCF) study, the safety and efficacy of oral supplementation of Fructosin® in fructose intolerance will be investigated.

The study participants will be informed about the nature and scope of the study during a preliminary examination (screening) and a declaration of consent will be obtained. In addition, it is determined whether fructose intolerance is present. This is determined by means of the aCPQ test. Subsequently, the patients fill out symptom questionnaires (IBS-SSS, IBS-QoL, 1-week symptom questionnaire).

After the eligibility check, a 14-day phase of monitoring and documentation of symptoms and complaints without taking Fructosin® (observation phase) takes place. At visit 1, the patients receive the Fructosin® capsules, which they take as needed, but no more than 2 x 3 times a day with fruit meals. The intake phase runs over a period of 28 days (4 weeks) during which the study participants observe and evaluate gastrointestinal symptoms with the help of the 1-weekly symptom questionnaire. In addition, the daily fructose consumption (fruit, fruit juices, smoothies) and the amount of Fructosin® capsules taken are documented in a diary.

ELIGIBILITY:
Inclusion Criteria:

* Positive result of the aCPQ test after 25 g fructose ingestion.
* Age: 18 - 80 years; 18 years of age must be completed and the legal capacity must be given.

Exclusion Criteria:

* Pregnancy and breastfeeding
* Congenital (hereditary) fructose intolerance
* Participation in a clinical trial in the past 4 weeks
* At the investigator's discretion: physical findings or previous illness for which a recommendation to take fructosin is not indicated or for which an assessment of the questionnaire by the patient is not possible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Test persons are recruited from the patient pool of the Clinical Department of Gastroenterology and Hepatology of the Medical University Clinic Graz. Fructose intolerance has been detected in these patients by means of aCPQ since March 2017. In addition, those affected will be approached through advertising measures and an aCPQ test for fructose intolerance determination will be carried out as part of the study. A detailed medical history will also be taken to check eligibility for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Safety of FRuctosin | 28 days
  Adverse events are recorded by the study participants by means of a diary and asked about by the study investigators at the end of the study (final visit).
  At the final visit, the subjects are asked about any changes in their health status. Any symptoms that occur that go beyond the symptoms of fructose intolerance are documented as adverse events (AE). All distinguishing features between adverse and serious adverse events, defined in accordance with the ICH/GCP guidelines, are queried and documented in the electronic case report form.
  AE are documented in source documents and include description, time period, treatment, intensity (1 mild, 2 moderate, 3 severe) and outcome (1 recovered, 2 recovered with limitation, 3 not yet recovered, 4 unknown), as well as severity (yes/no) and possible association (0 no association, 1 unlikely, 2 possible, 3 probable, 4 certain). The assessment of the association of AEs with the study medication is made by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Sciotec Diagnostic Technologies GmbH, Tulln, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No